CLINICAL TRIAL: NCT02089087
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose First-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CFZ533 in Healthy Subjects and Rheumatoid Arthritis Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Dose CFZ533 in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCFZ533X2101
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, RA, first-in-human, single ascending dose, safety, tolerability
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iscalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CFZ533 in healthy volunteers (Experimental): CFZ533 single dose in healthy volunteers
  Interventions: Biological: CFZ533
- CFZ533 in rheumatoid arthritis patients (Experimental): CFZ533 single dose in rheumatoid arthritis patients
  Interventions: Biological: CFZ533
- Placebo (Placebo Comparator): Placebo single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CFZ533 — Single dose at varying dosage levels depending on treatment assignment
  Arms: CFZ533 in healthy volunteers; CFZ533 in rheumatoid arthritis patients
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a first-in-human study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single intravenous and subcutaneous doses of CFZ533 in healthy subjects and intravenous doses in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This was a Healthy Volunteer only study originally, but after an amendment to protocol, rheumatoid arthritis patients will be starting 7-Mar-2014 and thus, the protocol is now registered.

ELIGIBILITY:
Inclusion Criteria (for healthy volunteers):

1. Healthy male and surgically sterilized or post-menopausal female subjects 18 to 55 years of age (for Cohort 9 only, subjects must be of Chinese descent)
2. Vital signs (systolic and diastolic blood pressure and pulse rate) should be within normal limits
3. Weight 50-150 kg and a body mass index (BMI) 18-32 kg/m2

Inclusion Criteria (for rheumatoid arthritis patients):

1. Healthy male and surgically sterilized or post-menopausal female subjects 18 to 55 years of age
2. Fulfilled 2010 ACR/EULAR classification criteria for RA per Investigator
3. Treatment with a stable oral RA treatment regimen for ≥ 4 weeks before randomization
4. Systemic corticosteroids allowed if on a stable dose (≤ 10 mg/day of prednisone or equivalent) ≥ 4 weeks prior to randomization
5. Subjects taking NSAIDs (COX-1 or COX-2 inhibitors) as part of their RA therapy must be on a stable dose for at least 4 weeks before randomization

Exclusion Criteria (for healthy volunteers):

1. History of hypersensitivity to vaccines, the study drug, or to drugs of similar chemical classes (i.e., biologic agents)
2. Abnormal hematology, coagulation or inflammatory lab results
3. History or evidence of tuberculosis.

Exclusion Criteria (for rheumatoid arthritis patients):

1. Use of anti-TNF or other biologics in previous 3 months
2. Any intra-articular injection therapy (e.g., corticosteroid, hyaluronan) required for treatment of acute RA flare within 4 weeks before randomization
3. Previous treatment with a B cell-depleting biologic agent or any other immunomodulatory biologic agent within 5 half-lives (experimental or approved)
4. Current treatment with cyclophosphamide
5. Autoimmune disease other than RA
6. Adult juvenile rheumatoid arthritis
7. RA functional status class IV according to the ACR 1991 revised criteria

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 7 months

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of CFZ533: Area Under the Plasma Concentration-time Curve (AUC) | 6 months
  The following PK parameters were determined from the plasma concentration time profile of CFZ533 using a non-compartmental method:
  AUCtau: Area under the plasma concentration-time curve from time zero to the end of the dosing interval
  AUClast: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
  AUCinf: Area under the plasma concentration-time curve from time zero to infinity
Plasma Pharmacokinetics (PK) of CFZ533: Observed Maximum Plasma Concentration Following Drug Administration (Cmax) | 6 months
Plasma Pharmacokinetics (PK) of CFZ533: Systemic Clearance from Plasma (CL) | 6 months
Plasma Pharmacokinetics (PK) of CFZ533: Apparent Volume of Distribution (Vss) | 6 months
CFZ533 immunogenicity | 6 months
  Determining the presence and measuring amount of anti-CFZ533 antibodies in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (5):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Duncansville, Pennsylvania
- Novartis Investigative Site, Taipei, Taiwan

REFERENCES:
- [Derived] Espie P, He Y, Koo P, Sickert D, Dupuy C, Chokote E, Schuler R, Mergentaler H, Ristov J, Milojevic J, Verles A, Groenewegen A, Auger A, Avrameas A, Rotte M, Colin L, Tomek CS, Hernandez-Illas M, Rush JS, Gergely P. First-in-human clinical trial to assess pharmacokinetics, pharmacodynamics, safety, and tolerability of iscalimab, an anti-CD40 monoclonal antibody. Am J Transplant. 2020 Feb;20(2):463-473. doi: 10.1111/ajt.15661. Epub 2019 Dec 6. PMID 31647605
- See also: Results for CCFZ533X2101 from the Novartis Trial Results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16987
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=283